CLINICAL TRIAL: NCT05404646
Title: Effects of Thoracic Mobility Versus Stretching Exercise Program on Pain, Range of Motion and Function in Patients of Cervical Radiculopathy.
Brief Title: Effects of Thoracic Mobility Versus Stretching Exercise Program in Patients of Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/22/0135 Iqra
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical radiculopathy; Thoracic spine; Thoracic mobilization; Stretching exercise
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Thoracic mobility exercises
  Interventions: Other: Thoracic mobility exercises with conventional physical therapy for cervical radiculopathy
- Group B (Experimental): Thoracic stretching exercises
  Interventions: Other: Thoracic stretching exercises with conventional physical therapy for cervical radiculopathy

INTERVENTIONS:
Other: Thoracic mobility exercises with conventional physical therapy for cervical radiculopathy — Thoracic mobility exercises These techniques include mobilization, manipulation and glides to check and treat the joints. Here, these techniques will be used to mobilize the thoracic spine. In this treatment mobility exercises (Unilateral posterior anterior, Central posterior anterior and transverse glides) + hot pack (10 min) + neck stretching (neck flexors, extensors, side benders) + cervical Traction will be given to patient. A total session time will be 45 min and thrice a week on alternate days for three weeks.
  Arms: Group A
Other: Thoracic stretching exercises with conventional physical therapy for cervical radiculopathy — Thoracic stretching exercises Thoracic stretching exercises. Thoracic stretching exercises are used to correct the musculature of thoracic region. In this treatment group stretching exercises (passive stretches and therapist facilitated exercises) +hot pack (10 min) +neck stretching (neck flexors, extensors, side benders) + tractions will be given to patient. A total of 45 min session thrice a week on alternate days for three weeks will be given. Only the eligible patients who fulfil the inclusion criteria will be included in the study.
  Arms: Group B

SUMMARY:
The study will be a randomized clinical trial with a sample size of 44 to determine the effects of thoracic mobility versus thoracic stretching exercises on pain, range of motion, and function in patients with cervical radiculopathy. Subjects will be enrolled according to inclusion-exclusion criteria. Patients will be divided into two groups, each with 22 patients. Group A will receive thoracic mobility exercises along with conventional physical therapy while group B will receive thoracic stretching exercises along with the conventional physical therapy protocol. The conventional physical therapy protocol will include a hot pack, neck Traction, and stretches. The session will be around 30 to 45 min for each patient with three sessions per week on alternate days. A total of Three weeks of treatment regime will be given to the patients and an assessment of patient's pain, range of motion, and function with the Numeric Pain Rating Scale (NPRS), goniometry and Neck Disability Index (NDI) will be done at the baseline, after the completion of treatment at three weeks and after six weeks to observe the long-term effects. will be analyzed by using SPSS version 25

DETAILED DESCRIPTION:
Cervical radiculopathy is characterized by neurological dysfunction caused by compression and inflammation of the spinal nerves or nerve roots of the cervical spine. The incidence and prevalence rate of cervical radiculopathy are unclear, and epidemiological data are limited.

Depending on the segments involved and the severity of neurological dysfunction, various signs and symptoms of cervical radiculopathy may manifest as neck and unilateral arm pain with numbness, weakness, or altered reflexes. Cervical spine radiculopathy is a disabling condition that has significant negative impacts on a person's mental health, physical functioning and social participation. It is a complex presentation, associated with increased dependence on healthcare systems, and poses a substantial challenge for clinicians and patients as it does not always respond to conventional therapies Symptoms of cervical radiculopathy may include neck and upper limb pain as well as neurological signs such as muscle weakness, disturbed sensation, and decreased reflex.

Patients with cervical radiculopathy demonstrated characteristics of sensory changes such as hypoesthesia (mechanical, thermal, and vibratory) and cold and pressure pain hypersensitivity. Conservative treatment, particularly physical therapy, is generally recommended as initial treatment for patients with cervical radiculopathy. It is found that vertebral mobilization and manipulation of the cervical spine were effective in improving pain, neck movement, and function in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria

* Both genders
* Age 25-55 years
* Unilateral cervical ridiculer pain.
* Chronicity of pain - 4 weeks minimum.
* Met wainner et al criteria (Slump test, Distraction test, ULTT)

Exclusion Criteria:

* • Fractures

  * Red Flags
  * Rheumatoid arthritis
  * Neurologic deficit
  * Injury to spinal cord
  * Tumor
  * Circulatory disturbances

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3rd Week
  The Numeric Pain Rating Scale (NPRS) is a popular method to assess pain. The Numeric Pain Rating Scale (NPRS), asks the patient to quantify their pain on scale from 0 to 10 using whole Arabic numbers. On this 0 refers the no pain and 10 refers the highest pain.
Neck Disability index | 3rd Week
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50
Range of Motion | 3rd Week
  The science of measuring the joint ranges in each plane of the joint is called goniometry. Goniometry is a device that measures an angle or permits the rotation of an object to a definite position. Neck flexion, extension, side bending will be assessed through it

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- District Head Quarter Bahawalnagar, Bahāwalnagar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang KC, Lee HS, Lee JH. Cervical Radiculopathy Focus on Characteristics and Differential Diagnosis. Asian Spine J. 2020 Dec;14(6):921-930. doi: 10.31616/asj.2020.0647. Epub 2020 Dec 22. PMID 33373515
- [Background] Mansfield M, Smith T, Spahr N, Thacker M. Cervical spine radiculopathy epidemiology: A systematic review. Musculoskeletal Care. 2020 Dec;18(4):555-567. doi: 10.1002/msc.1498. Epub 2020 Jul 25. PMID 32710604
- [Background] Alshami AM, Bamhair DA. Effect of manual therapy with exercise in patients with chronic cervical radiculopathy: a randomized clinical trial. Trials. 2021 Oct 18;22(1):716. doi: 10.1186/s13063-021-05690-y. PMID 34663421
- [Background] Liang L, Feng M, Cui X, Zhou S, Yin X, Wang X, Yang M, Liu C, Xie R, Zhu L, Yu J, Wei X. The effect of exercise on cervical radiculopathy: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Nov;98(45):e17733. doi: 10.1097/MD.0000000000017733. PMID 31702624
- [Background] Hassan F, Osama M, Ghafoor A, Yaqoob MF. Effects of oscillatory mobilization as compared to sustained stretch mobilization in the management of cervical radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(1):153-158. doi: 10.3233/BMR-170914. PMID 31127753
- [Background] Heneghan NR, Lokhaug SM, Tyros I, Longvastol S, Rushton A. Clinical reasoning framework for thoracic spine exercise prescription in sport: a systematic review and narrative synthesis. BMJ Open Sport Exerc Med. 2020 Mar 29;6(1):e000713. doi: 10.1136/bmjsem-2019-000713. eCollection 2020. PMID 32341799
- [Background] Ali AA, Sheikh N, Chughani V, Hussain A, Rafique M, Ismail M, et al. Comparision of Effectiveness of Isometric and Stretching Exercise in Pain Management among the Forward Head Posture Patients. Indian Journal of Physiotherapy & Occupational Therapy. 2021;15(2).
- [Background] Young IA, Pozzi F, Dunning J, Linkonis R, Michener LA. Immediate and Short-term Effects of Thoracic Spine Manipulation in Patients With Cervical Radiculopathy: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2019 May;49(5):299-309. doi: 10.2519/jospt.2019.8150. Epub 2019 Apr 25. PMID 31021691
- [Background] Langevin P, Desmeules F, Lamothe M, Robitaille S, Roy JS. Comparison of 2 manual therapy and exercise protocols for cervical radiculopathy: a randomized clinical trial evaluating short-term effects. J Orthop Sports Phys Ther. 2015 Jan;45(1):4-17. doi: 10.2519/jospt.2015.5211. PMID 25420010
- [Background] Borrella-Andres S, Marques-Garcia I, Lucha-Lopez MO, Fanlo-Mazas P, Hernandez-Secorun M, Perez-Bellmunt A, Tricas-Moreno JM, Hidalgo-Garcia C. Manual Therapy as a Management of Cervical Radiculopathy: A Systematic Review. Biomed Res Int. 2021 Jun 3;2021:9936981. doi: 10.1155/2021/9936981. eCollection 2021. PMID 34189141